CLINICAL TRIAL: NCT06238661
Title: Prostate Cancer Screening With PSA, Risk Calculator and Multiparametric MRI: a Pilot Study
Brief Title: Prostate Cancer Screening: a Pilot Study
Acronym: ProScreenMRI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Collaborators: San Luigi Gonzaga Hospital (Other); Epidemiology and Screening Unit - CPO, Turin, Italy (Unknown); ASL TO5 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ProScreenMRI
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PSA; Risk Calculator; Magnetic Resonance Imaging; Prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with PSA ≥ 3 ng/ml (Experimental): * Urologic examination
  * Risk calculation (ERSPC no.6)
  * Magnetic resonance imaging
  * (optional) biopsy
  Interventions: Diagnostic Test: Urology visit with Risk Calculator and MRI

INTERVENTIONS:
Diagnostic Test: Urology visit with Risk Calculator and MRI — Patients with PSA ≥3 ng/ml will undergo urology visit with risk calculator and MRI assessment of the prostate

SUMMARY:
Prostate Cancer (PCa) is the second most frequently diagnosed tumour and the third most lethal among men in Europe. The lack of precise tools and examinations to precisely diagnose PCa has caused overtreatment of indolent and low-aggressive PCa, while in some other cases, with aggressive disease, diagnosis and treatment are dangerously delayed because cancer could be potentially missed. The present trial aims to study a new pathway to early diagnose PCa with Magnetic Resonance Imaging (MRI) to identify men who will not need treatment and those who will benefit from radical treatment, thus improving disease control and quality of life.

DETAILED DESCRIPTION:
Men aged 55-65 years with neither previous biopsy nor prostate diseases will be invited in the screening protocol and will perform an initial PSA test. Those cases with PSA ≥ 3 ng/ml will be invited to undergo a urologic examination with computed risk assessment and an MRI, which is a non-invasive test with high positive and negative predictive value in identifying clinically significant prostate cancer. Then, only men with medium-high risk of harbouring clinically significant prostate cancer will be invited to undergo a prostate biopsy to indentify cancer presence and its aggressiveness.

ELIGIBILITY:
Inclusion Criteria:

* age between 55-65 years;
* asymptomatic or paucisymptomatic from a urological point of view;
* no previous prostate biopsy;
* living in the ASL TO5 (Piedmont, Italy);
* signed written informed consent.

Exclusion Criteria:

* positive oncologic anamnesis for prostate cancer;
* previous biopsy or prostate surgery;
* previous radiotherapy of the pelvis;
* any contraindication to MRI examination;
* claustrophobic or uncollaborative subjects.

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4500 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer (Gleason Group ≥2) | 24 months
  No. of detected clinically significant prostate cancer with Gleason Group ≥ 2 over the total no. of men enrolled in the trial
Comparison of the detection rate of clinically significant prostate cancer with and without screening | 24 months
  No. of detected clinically significant prostate cancer with Gleason Group ≥ 2 over the total no. of men enrolled in the trial compared to the same proportion of men calculated in the 2-year period before the introduction of the screening protocol
Verify that the detection rate of clinically significant prostate cancer with the screening strategy is not inferior to that of the Italian cohort in the ERSPC study | 24 months
  No. of detected clinically significant prostate cancer with Gleason Group ≥ 2 over the total no. of men enrolled in the trial compared to the same proportion of men included in the Italian cohort of the ERSPC study screened using PSA only

SECONDARY OUTCOMES:
Changes in number of biopsy procedures | 24 months
  Estimation of the number of biopsy that could be avoided using the new screening strategy compared to the use of PSA only.
Assessment of positive and negative predictive values | 24 months
  Definition of positive and negative predictive values of the proposed screening strategy and comparison with those obtained in the ERSPC screening study with PSA only

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Regge, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia, Candiolo, Italy, Italy

IPD SHARING:
Plan to Share IPD: No